CLINICAL TRIAL: NCT04013867
Title: Identification of the Best Self-questionnaire to Diagnose Depression in Patients With Psoriasis
Brief Title: Identification of the Best Self-questionnaire to Diagnose Depression in Patients With Psoriasis (DePsoVal)
Acronym: DePsoVal
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2019 LAURON; 2019-A01119-48 (Other: ANSM)
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Psoriasis; Depression
Keywords: psoriasis; depression; validation; self-questionnaire
MeSH Terms: conditions — Psoriasis; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prevalence of depression shows great heterogeneity in patients with psoriasis. This could be explained by the psychometric properties of the questionnaires assessing depressive symptoms: these tests have not been developed in a context of dermatosis. The complaints and symptoms associated with psoriasis can be misidentified by questionnaires as a manifestation of depressive symptomatology and may overestimate depressive symptoms.

In other diseases such as asthma and rheumatoid arthritis, tools have been validated specifically to take into account these symptoms.

The purpose of this study is to validate and compare assessment tools for depression in patients with psoriasis.

DETAILED DESCRIPTION:
The study does not modify the management of patients. Patients will be contacted by phone. The protocol, the modalities and the objectives of the study will be presented during a first telephone interview. A second telephone interview will be scheduled with the patient 3 days later for the collection of his informed consent, if he agrees to participate, and the completion of the questionnaires of the study. The online questionnaires will be sent by email during this call.

1. Telephone interview (5 minutes) Presentation of the study. Schedule a telephone appointment 3 days later.
2. Telephone interview (10 minutes) Collection of consent. Sociodemographic questionnaire: sex, age, marital status, level of education Medical questionnaire including the consumption of tobacco and alcohol, the collection of current treatments, their indications and their start dates.

   Semi-directed telephone interview to identify the presence of depressive or dysthymic disorders (MINI).
3. mailing of the self-questionnaires (20 to 30 minutes) Medical questionnaire: duration of psoriasis, simplified index of psoriasis, presence of pruritus, pain EVA (cutaneous and articular), fatigue.

   Self-questionnaires BDI, PHQ9, IDS, QIDS, HADS assessing the intensity of depressive symptoms.
4. Retest (10 minutes) Some patients will be offered to re-fill the self-questionnaires assessing the intensity of depressive symptoms 15 days after completion of the survey. All participants selected for the retest will not complete all questionnaires again: the questionnaires will be distributed among the patients. The retest requires 50 patients who declare themselves stable (identified by one item) for each questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Major patient, male or female, with psoriasis, less than 65 years old, followed up in the dermatology or rheumatology departments of the University Hospital of Clermont-Ferrand.
* Able to mentally and linguistically answer the proposed questionnaires.
* Can fill out online questionnaires from his home.
* Affiliated with Social Security.

Exclusion Criteria:

* Major incapable patient
* Refusal of participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with psoriasis
Sampling Method: Non-Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance in term of specificity of self-questionnaires assessing depression in relation to the diagnosis made during the interview using the MINI (Mini International neuropsychiatric Interview) | Day 7
  Comparison of specificity between each self-questionnaires (PHQ9- Patient health Questionnaire, BDI - Beck Depression Inventory, HADS, Hospital Anxiety and Depression Scale-Depression, IDS, Inventory of Depressive Symptomatology ). Threshold values will be determined with the ROC curves according to presence of depression or not (identified during with the MINI).
Diagnostic performance in term of positive predictive value of self-questionnaires assessing depression in relation to the diagnosis made during the interview using the MINI (Mini International neuropsychiatric Interview) | Day 7
  Comparison of positive predictive values according to threshold values between each self-questionnaires (PHQ9- Patient health Questionnaire, BDI - Beck Depression Inventory, HADS, Hospital Anxiety and Depression Scale-Depression, IDS, Inventory of Depressive Symptomatology ). Threshold values will be determined with the ROC curves according to presence of depression or not (identified during with the MINI).
Diagnostic performance in term of sensitivity of self-questionnaires assessing depression in relation to the diagnosis made during the interview using the MINI (Mini International neuropsychiatric Interview) | Day 7
  Comparison of sensitivity between each self-questionnaires (PHQ9- Patient health Questionnaire, BDI - Beck Depression Inventory, HADS, Hospital Anxiety and Depression Scale-Depression, IDS, Inventory of Depressive Symptomatology ). Threshold values will be determined with the ROC curves according to presence of depression or not (identified during with the MINI).
Diagnostic performance in term of negative predictive value of self-questionnaires assessing depression in relation to the diagnosis made during the interview using the MINI (Mini International neuropsychiatric Interview) | Day 7
  Comparison of negative predictive values according to threshold values between each self-questionnaires (PHQ9- Patient health Questionnaire, BDI - Beck Depression Inventory, HADS, Hospital Anxiety and Depression Scale-Depression, IDS, Inventory of Depressive Symptomatology ). Threshold values will be determined with the ROC curves according to presence of depression or not (identified during with the MINI).

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Lauron, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France